CLINICAL TRIAL: NCT05921175
Title: A Pilot Study on the Cumulative Effects of Transcutaneous Spinal Cord Stimulation (tSCS) With Robotic Gait Training in Trunk Muscle Activity and Walking Index in Chronic Spinal Cord Injury
Brief Title: tSCS + EksoGT in SCI Patients
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National University Hospital, Singapore (Other)
Collaborators: Alexandra Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 2023/00350
Record Dates: First submitted 2023-06-19; First posted 2023-06-27 (Actual); Last update posted 2024-08-16 (Actual); Status verified 2024-08

CONDITIONS: Spinal Cord Injury
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Intervention Model Description: This is a prospective single-arm crossover study in participants with incomplete chronic traumatic spinal cord paraplegia.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- RGT+ conventional physiotherapy (Active Comparator): 16 sessions of robotic gait training (RGT) + conventional physiotherapy in 8-10 weeks
  Interventions: Device: RGT+ conventional physiotherapy
- RGT+ tSCS + conventional physiotherapy (Experimental): Phase 2: 16 sessions of RGT training + transcutaneous electrical stimulation (tSCS) + functional training in 8-10 weeks.
  Interventions: Device: RGT+ tSCS + conventional physiotherap

INTERVENTIONS:
Device: RGT+ tSCS + conventional physiotherap — Subject will undergo 16 sessions of robotic gait training (RGT) + tSCS+ conventional physiotherapy in 8-10 weeks. Subject will walk with EksoGT for gait training during RGT training. Components of conventional physiotherapy will include upper/lower limb ergometry and strength training as prescribed by the attending physiotherapist based on their assessment. During tSCS, cathodes will be placed on the T11 and L1 spinous process. Reference/Ground electrodes placed over the ASIS It will be on biphasic mode with an overlap frequency of 10kHz, Burst Frequency of 30Hz, Pulse width of 1ms. Stimulation intensity ranges from 5-100 mA and will be adjusted according to the patient's response. The tSCS stimulation duration for each session will be 45 minutes in conjunction with the RGT training.
  Arms: RGT+ tSCS + conventional physiotherapy
Device: RGT+ conventional physiotherapy — Subject will undergo 16 sessions of robotic gait training (RGT) + conventional physiotherapy in 8-10 weeks. Subject will walk with EksoGT for gait training during RGT training. Components of conventional physiotherapy will include upper/lower limb ergometry and strength training as prescribed by the attending physiotherapist based on their assessment.
  Arms: RGT+ conventional physiotherapy

SUMMARY:
This study is aimed to evaluate whether transcutaneous spinal cord stimulation (tSCS) can augment robotic gait training (RGT) to improve functional mobility in participants with chronic paraplegia. It also evaluate the impact of the tSCS+RGT on health-related quality of life (HRQOL), compared to RGT alone.

This is a prospective single-arm crossover study in participants with incomplete chronic traumatic spinal cord paraplegia. 6 subjects will be recruited. The intervention includes Phase 1 of training which consists of 16 sessions of robotic gait training (RGT) + conventional physiotherapy in 8-10 weeks, and Phase 2 of training which consists of 16 sessions of RGT training + tSCS + conventional physiotherapy in 8-10 weeks.

Outcome measures including mobility function assessment and neuromuscular assessment will be collected at Baseline, Post-Phase 1 and Post-Phase 2. A satisfaction survey on the intervention "RGT training + tSCS + conventional physiotherapy" will be performed at week-18 assessment.

DETAILED DESCRIPTION:
This study is aimed to evaluate whether transcutaneous spinal cord stimulation (tSCS) can augment robotic gait training (RGT) to improve functional mobility in participants with chronic paraplegia. It also evaluate the impact of the tSCS+RGT on health-related quality of life (HRQOL), compared to RGT alone.

This is a prospective single-arm crossover study in participants with incomplete chronic traumatic spinal cord paraplegia. 6 subjects will be recruited. Once subject is identified to be eligible for the study and is agreeable to participate into the study, he/she will undergo Phase 1 of training which consists of 16 sessions of robotic gait training (RGT) + conventional physiotherapy in 8-10 weeks. After a 1-week washout period, subject will undergo Phase 2 of training which consists of 16 sessions of RGT training + tSCS + conventional physiotherapy in 8-10 weeks.

Subject will walk with EksoGT for gait training during RGT training. Components of conventional physiotherapy will include upper/lower limb ergometry and strength training as prescribed by the attending physiotherapist based on their assessment. During tSCS, cathodes will be placed on the T11 and L1 spinous process. Reference/Ground electrodes placed over the ASIS It will be on biphasic mode with an overlap frequency of 10kHz, Burst Frequency of 30Hz, Pulse width of 1ms. Stimulation intensity ranges from 5-100 mA and will be adjusted according to the patient's response. The tSCS stimulation duration for each session will be 45 minutes in conjunction with the RGT training.

Outcome measures including mobility function assessment and neuromuscular assessment will be collected at Baseline (within 1 week before the starting of Phase 1 of training), Post-Phase 1 (within 1 week after Phase 1 of training) and Post-Phase 2 (within 1 week after Phase 2 of training).

A satisfaction survey on the intervention "RGT training + tSCS + conventional physiotherapy" will be performed at week-18 assessment.

ELIGIBILITY:
Inclusion Criteria:

1. Between 6 months to 5 years from the diagnosis of the traumatic SCI and who are not walking independently;
2. Age between 21 to 65 years old;
3. Incomplete spinal cord injury: ASIA Impairment Scale (AIS) Grade: B-D;
4. Spinal cord injury level: T1- L1;
5. SCI-TCT Score > 13;
6. Capable of providing an informed consent;
7. Cleared by Neurosurgeons/ Orthopeadic Surgeons for tSCS;
8. Meets prerequisites for Ekso wearable robotic exoskeleton training.

Exclusion Criteria:

1. Participant has uncontrolled cardiopulmonary disease or cardiac symptoms as determined by the investigator;
2. Participant has any unstable or significant medical condition that is likely to interfere with study procedures or likely to confound performance and outcomes like uncontrolled neuropathic pain, depression, severe cognitive impairment;
3. Unstable or uncontrolled autonomic dysreflexia;
4. Requires ventilator support;
5. Spasms that limit the ability of the subjects to participate in the study training as determined by the investigator;
6. Skin conditions that limit the application of tSCS electrodes;
7. Active implanted medical devices that may be affected by tSCS;
8. Pregnant, planning to become pregnant or breastfeeding;
9. Concurrent participation in another drug or device trial that may interfere with this study;
10. Participated in wearable exoskeleton training within the last 3 months prior to enrolment.
11. Peripheral nerve injury or significant Lumbar Radiculopathy

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Estimated)
Dates: Start 2024-11 (Estimated); Primary Completion 2026-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Spinal Cord Injury - Trunk Control Test (SCI-TCT) | Week 0
  It measures 4 simple aspect of trunk movement: 1) rolling to weak side; 2) rolling to strong side; 3) balance in sitting position; 4) sit up from lying down. The final score ranges from 0 (minimum) to 100 (maximum, indicating better performance)
Spinal Cord Injury - Trunk Control Test (SCI-TCT) | Week 8
  It measures 4 simple aspect of trunk movement: 1) rolling to weak side; 2) rolling to strong side; 3) balance in sitting position; 4) sit up from lying down. The final score ranges from 0 (minimum) to 100 (maximum, indicating better performance)
Spinal Cord Injury - Trunk Control Test (SCI-TCT) | Week 17
  It measures 4 simple aspect of trunk movement: 1) rolling to weak side; 2) rolling to strong side; 3) balance in sitting position; 4) sit up from lying down. The final score ranges from 0 (minimum) to 100 (maximum, indicating better performance)
Walking Index in Spinal Cord Injury-II (WISCI-II) | Week 0
  It is an ordinal scale of 20 items assessing the amount of physical assistance needed, as well as device required, for walking following paralysis that results from spinal cord injury. Final score ranges from 0 (minimum) to 20 (maximum, indicating better performance).
Walking Index in Spinal Cord Injury-II (WISCI-II) | Week 8
  It is an ordinal scale of 20 items assessing the amount of physical assistance needed, as well as device required, for walking following paralysis that results from spinal cord injury. Final score ranges from 0 (minimum) to 20 (maximum, indicating better performance).
Walking Index in Spinal Cord Injury-II (WISCI-II) | Week 17
  It is an ordinal scale of 20 items assessing the amount of physical assistance needed, as well as device required, for walking following paralysis that results from spinal cord injury. Final score ranges from 0 (minimum) to 20 (maximum, indicating better performance).
10-Meter Walk Test (10MWT) | Week 0
  It measures walking speed when subject walks at comfortable speed, covered in the distance of 10 meters. Higher result indicates higher walking speed/better performance.
10-Meter Walk Test (10MWT) | Week 8
  It measures walking speed when subject walks at comfortable speed, covered in the distance of 10 meters. Higher result indicates higher walking speed/better performance.
10-Meter Walk Test (10MWT) | Week 17
  It measures walking speed when subject walks at comfortable speed, covered in the distance of 10 meters. Higher result indicates higher walking speed/better performance.
Central motor conduction time (CMCT) | Week 0
  Measured by transcranial magnetic stimulation (TMS). It is calculated by subtracting the peripheral conduction time (PMCT) from motor evoked potential (MEP) latency elicited by TMS to the motor cortex. Higher results indicates longer central motor conduction time and poor performance.
Central motor conduction time (CMCT) | Week 8
  Measured by transcranial magnetic stimulation (TMS). It is calculated by subtracting the peripheral conduction time (PMCT) from motor evoked potential (MEP) latency elicited by TMS to the motor cortex. Higher results indicates longer central motor conduction time and poor performance.
Central motor conduction time (CMCT) | Week 17
  Measured by transcranial magnetic stimulation (TMS). It is calculated by subtracting the peripheral conduction time (PMCT) from motor evoked potential (MEP) latency elicited by TMS to the motor cortex. Higher results indicates longer central motor conduction time and poor performance.
International standards for Neurological Classification of SCI (ISNCSCI) | Week 0
  The test is to define and describe the extent and severity of a patient's spinal cord injury. The patient's grade is based on how much sensation he or she can feel at multiple points on the body, as well as tests of motor function. The results ranged from A (worst- complete lack of motor and sensory function below the level of injury) to E (best, all neurologic function has returned)
International standards for Neurological Classification of SCI (ISNCSCI) | Week 8
  The test is to define and describe the extent and severity of a patient's spinal cord injury. The patient's grade is based on how much sensation he or she can feel at multiple points on the body, as well as tests of motor function. The results ranged from A (worst- complete lack of motor and sensory function below the level of injury) to E (best, all neurologic function has returned)
International standards for Neurological Classification of SCI (ISNCSCI) | Week 17
  The test is to define and describe the extent and severity of a patient's spinal cord injury. The patient's grade is based on how much sensation he or she can feel at multiple points on the body, as well as tests of motor function. The results ranged from A (worst- complete lack of motor and sensory function below the level of injury) to E (best, all neurologic function has returned)

SECONDARY OUTCOMES:
EQ5D | Week 0
  EQ5D is an instrument which evaluates the generic quality of life developed in Europe and widely used. It has one question for each of the five dimensions that include mobility, self-care, usual activities, pain/discomfort, and anxiety/depression, each dimension scored from 1 to 5, the higher score indicates worse performance.
EQ5D | Week 8
  EQ5D is an instrument which evaluates the generic quality of life developed in Europe and widely used. It has one question for each of the five dimensions that include mobility, self-care, usual activities, pain/discomfort, and anxiety/depression, each dimension scored from 1 to 5, the higher score indicates worse performance.
EQ5D | Week 17
  EQ5D is an instrument which evaluates the generic quality of life developed in Europe and widely used. It has one question for each of the five dimensions that include mobility, self-care, usual activities, pain/discomfort, and anxiety/depression, each dimension scored from 1 to 5, the higher score indicates worse performance.
Modified Tardieu Scale | Week 0
  Modified Tardieu Scale is to measure if there is spasticity present in a person's muscle and its response to movement. It will be measured for Quadriceps, Hamstrings, Gastrocnemius. A large difference between R1 and R2 suggests a large dynamic component with a greater capacity for change or improvement. A small difference between R1 and R2 suggests a predominantly fixed contracture in the muscle with a poorer capacity for change
Modified Tardieu Scale | Week 8
  Modified Tardieu Scale is to measure if there is spasticity present in a person's muscle and its response to movement. It will be measured for Quadriceps, Hamstrings, Gastrocnemius. A large difference between R1 and R2 suggests a large dynamic component with a greater capacity for change or improvement. A small difference between R1 and R2 suggests a predominantly fixed contracture in the muscle with a poorer capacity for change
Modified Tardieu Scale | Week 17
  Modified Tardieu Scale is to measure if there is spasticity present in a person's muscle and its response to movement. It will be measured for Quadriceps, Hamstrings, Gastrocnemius. A large difference between R1 and R2 suggests a large dynamic component with a greater capacity for change or improvement. A small difference between R1 and R2 suggests a predominantly fixed contracture in the muscle with a poorer capacity for change
EMG measurement | Week 0
  EMG signals from bilateral Quadriceps, Tibialis Anterior, Gastrocnemius, Rectus Abdominis will be recorded for about 10 seconds. Root-Mean-Square (RMS) of the EMG signals will be calculated.
EMG measurement | Week 8
  EMG signals from bilateral Quadriceps, Tibialis Anterior, Gastrocnemius, Rectus Abdominis will be recorded for about 10 seconds. Root-Mean-Square (RMS) of the EMG signals will be calculated.
EMG measurement | Week 17
  EMG signals from bilateral Quadriceps, Tibialis Anterior, Gastrocnemius, Rectus Abdominis will be recorded for about 10 seconds. Root-Mean-Square (RMS) of the EMG signals will be calculated.

CONTACTS AND LOCATIONS:
Overall Officials: Gobinathan Chandran, MBBS, Principal Investigator — National University Hospital, Singapore
Locations (1):
- Alexandra Hospital, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No